CLINICAL TRIAL: NCT07251062
Title: A Phase II/III Study to Evaluate the Efficacy and Safety of SYS6010 in Combination With SG001 With or Without 5-FU/Capecitabine in Subjects With First-Line Advanced/Metastatic Esophageal Squamous Cell Carcinoma.
Brief Title: A Study of SYS6010, Enlonstobart, and Chemotherapy for First-Line Treatment of Esophageal Squamous Cell Carcinoma.
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYS6010-016
Record Dates: First submitted 2025-11-13; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Intervention Model Description: This is a Phase II/III study. Phase II study comprises a safety lead-in stage, a dose expansion stage, and a randomized treatment stage. The Phsae III study is randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Phase II (Safety lead-in stage) : SYS6010+SG001+physician's choice(Capecitabine or 5-FU ) (Experimental)
  Interventions: Drug: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU)
- Phase II (dose expansion stage): SYS6010+SG001+physician's choice (Capecitabine or 5-FU) (Experimental): Upon completion of the safety evaluation and confirmation of tolerability for a dose cohort in the safety run-in phase, expansion of that cohort may be initiated, with plans to expand 1-2 dose cohorts.
  Interventions: Drug: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU)
- Phase II(randomized Controlled stage): SYS6010+SG001+ physician's choice (Capecitabine or 5-FU) (Experimental)
  Interventions: Drug: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU)
- PhaseII(randomized treatment stage): physician's choice of SOC (Active Comparator)
  Interventions: Drug: Investigator's choice of SOC
- Phase II(randomized controlled stage): SYS6010+SG001 (Experimental)
  Interventions: Drug: SYS6010+SG001
- Phase III: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU) (Active Comparator)
  Interventions: Drug: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU)
- Phase III: physician's choice of SOC (Active Comparator)
  Interventions: Drug: Investigator's choice of SOC

INTERVENTIONS:
Drug: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU) — SYS6010 is an antibody conjugate drug (ADC), composed of one anti-EGFR monoclonal antibody coupled to one JS1 via an enzyme specific linker.
  SG001 is a recombinant, fully human, anti-PD-1 monoclonal antibody. Capecitabine: Capecitabine is for oral administration. 5-FU: Administration at the conventional dosage.
  Other Names: SG001: Enlonstobart
  Arms: Phase II (Safety lead-in stage) : SYS6010+SG001+physician's choice(Capecitabine or 5-FU ); Phase II (dose expansion stage): SYS6010+SG001+physician's choice (Capecitabine or 5-FU); Phase II(randomized Controlled stage): SYS6010+SG001+ physician's choice (Capecitabine or 5-FU); Phase III: SYS6010+SG001+ physician's choice (Capecitabine or 5-FU)
Drug: Investigator's choice of SOC — 1. Camrelizumab + Cisplatin + Paclitaxel
  2. Tislelizumab + Cisplatin + Paclitaxel
  3. Tislelizumab + Cisplatin + 5-FU/Capecitabine
  Arms: Phase III: physician's choice of SOC; PhaseII(randomized treatment stage): physician's choice of SOC
Drug: SYS6010+SG001 — SYS6010 is an antibody conjugate drug (ADC), composed of one anti-EGFR monoclonal antibody coupled to one JS1 via an enzyme specific linker.
  SG001 is a recombinant, fully human, anti-PD-1 monoclonal antibody.
  Arms: Phase II(randomized controlled stage): SYS6010+SG001

SUMMARY:
This is a multicenter phase 2/3 clinical study to evaluate the efficacy and safety of SYS6010 plus SG001±5-FU/Capecitabine as first-line treatment, in patients with advanced/metastatic esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Phase II study comprises a safety lead-in stage, a dose expansion stage, and a randomized treatment stage. The Phsae III study is randomized controlled trial.

Phase II (safety lead-in stage): the safety lead-in stage employs a 3+3 design. It aims to evaluate the safety and tolerability of combination therapy-comprising capecitabine/5-FU administered at a descending dose level starting from DL0 alongside fixed doses of SYS6010 and SG001-in previously untreated patients with unresectable locally advanced or metastatic ESCC. The primary objectives are to determine the Maximum Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D).

Phase II (dose expansion stage): Upon completion of the safety evaluation and confirmation of tolerability for a dose cohort in the safety lead-in phase, expansion of that cohort may be initiated, with plans to expand 1-2 dose cohorts.

Phase II (randomized treatment stage): Upon determination of the RP2D based on prior data, a randomized controlled study will be conducted in a first-line advanced/metastatic esophageal squamous cell carcinoma (ESCC) patient population. Patients will be randomly assigned to three arms: Arm 1: SYS6010+SG001+ capecitabine/5-FU; arm2: investigator's choice of SOC; arm3: SYS6010+SG001.

Phase III is a randomized, controlled, open-label, multicenter study designed to evaluate the efficacy of SYS6010+SG001+capecitabine/5-FU versus investigator's choice of treatment as first-line therapy for advanced/metastatic esophageal squamous cell carcinoma. The Phase III trial design will be finalized based on Phase II results. The preliminary plan is to randomized patients in a 1:1 ratio to either the investigational arm or the control arm. Investigational arm: SYS6010+SG001+capecitabine/5-FU; control arm: investigator's choice of SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and voluntarily sign the written ICF;
2. Age 18-75 (inclusive) years, male or female;
3. With histologically/cytologically confirmed esophageal squamous cell carcinoma that is either locally advanced unresectable or metastatic, with no prior systemic antitumor therapy administered for the recurrent/metastatic disease setting. Have at least one measurable lesion that meets the RECIST v 1.1 criteria at baseline;
4. Eastern Cooperative Oncology Group (ECOG) performance status score: 0-1;
5. Life expectancy ≥ 3 months;

Exclusion Criteria:

1. Prior treatment involving topoisomerase I inhibitors (including ADC drugs that contain topoisomerase I inhibitors as toxins);
2. Prior treatment with immune checkpoint inhibitors or other agents targeting T-cell co-stimulatory/co-inhibitory pathways (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-CD137 antibodies)
3. With a history of ≥Grade 3 allergic reactions to monoclonal antibodies, or with known hypersensitivity or intolerance to SYS6010, SG001, paclitaxel, carboplatin, cisplatin, fluorouracil, or any of their excipients;
4. With dihydropyrimidine dehydrogenase (DPD) deficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 737 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
PhaseII(safety leadrun-in stage): DLT; Description: Dose-limiting toxicity | 28 days
  Dose-limiting toxicity
PhaseII(safety run-inlead-in stage): AE | From the signing of the informed consent form until 90 days after the last dose.
  The incidence and severity of Adverse events
PhaseII(safety leadrun-in stage): MTD; | After phase II saftysafety run-inlead-in stage and dose expansion stage. Approximately 4 months.
  Maximum tolerated dose
PhaseII(safety run-inlead-in stage): RP2D | After phase II saftysafety run-inlead-in stage and dose expansion stage. Approximately 4 months.
  Recommended Phase II dose
PhaseII(Randomized treatment stage): ORR per RECIST v1.1 | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years.
  Objective response rate
PhaseIII: PFS-ICR | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years
  PFS assessed by independent review committee
PhaseIII: OS; | Through study completion, up to approximately 5 year.
  Overall survival

SECONDARY OUTCOMES:
Phase II: DOR per RECIST 1.1; | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years
  Duration of response.
Phase II: DCR per RECIST 1.1; | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years
  Disease of controll
Phase II:PFS per RECIST 1.1 | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years
  Progression free survival
Phase II:OS | Through study completion, up to approximately 5 year
  Overall survival
Phase II: Serum concentrations of toxin-bound antibodies, total antibodies, and JS-1 following single and multiple doses of SYS6010 | From first dose of treatment to 30 days after the last dose of treatment.
  Serum concentrations of toxin-bound antibodies, total antibodies, and JS-1 following single and multiple doses of SYS6010
Phase II: plasma concentration of SG001 following single and multiple doses of SG001; | From first dose of treatment to 30 days after the last dose of treatment.
  Plasma concentration of SG001 following single and multiple doses of SG001
Phase II: EGFR protein expression and PD-L1 protein expression; | From first dose of treatment to 30 days after the last dose of treatment.
  EGFR protein expression and PD-L1 protein expression;
Phase II: The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SYS6010. | From first dose of treatment to 30 days after the last dose of treatment.
  The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SYS6010.
Phase II: The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SG001; | From first dose of treatment to 30 days after the last dose of treatment.
  The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SG001.
Phase III: DOR-IRC per RECIST 1.1 | Weeks 8, 12, 18, every 6 weeks within 48 weeks, and every 12 weeks thereafter, until the end of the study
  Duration of response assessed by independent review committee
Phase III: DCR-IRC per RECIST 1.1; | Weeks 8, 12, 18, every 6 weeks within 48 weeks, and every 12
  Disease of controll assessed by independent review committee.
Phase III:PFS per RECIST 1.1; | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years.
  Progression free survival
Phase III:ORR-IRC; | From date of randomization until the date of ﬁrst documented progression or date of death from any cause, whichever came ﬁrst, assessed up to 5 years.
  Objective response rate assessed by independent review committee
Phase III: AE; | From first dose of treatment to 90 days after the last dose of treatment.
  Incidence and severity of adverse events
Phase III: Serum concentrations of toxin-bound antibodies, total antibodies, and JS-1 following single and multiple doses of SYS6010; | From first dose of treatment to 30 days after the last dose of treatment.
  Serum concentrations of toxin-bound antibodies, total antibodies, and JS-1 following single and multiple doses of SYS6010
Phase III: plasma concentration of SG001 following single and multiple doses of SG001 | From first dose of treatment to 30 days after the last dose of treatment.From first dose of treatment to 30 days after the last dose of treatment.
  Plasma concentration of SG001 following single and multiple doses of SG001
Phase III: EGFR protein expression and PD-L1 protein expression | From first dose of treatment to 30 days after the last dose of treatment.
  EGFR protein expression and PD-L1 protein expression
Phase III: The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SYS6010 . | From first dose of treatment to 30 days after the last dose of treatment.
  The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SYS6010.
The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SG001 | From first dose of treatment to 30 days after the last dose of treatment
  The incidence and titer of anti-drug antibodies (ADA), as well as the incidence of neutralizing antibodies (NAb) (if applicable), for SG001